CLINICAL TRIAL: NCT02960425
Title: Randomized, Double-blind, Placebo-controlled, Short Term Trial of DelivraTM Livsport Preworkout Cream for Improved Power Output and Reduction of Muscle Fatigue During Resistant Training
Brief Title: Delivra Topical Creatine for Improving Muscular Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 16-145a
Record Dates: First submitted 2016-10-30; First posted 2016-11-09 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HI Delivra TM Livsport preworkout cream (Experimental): 7 mL topical creatine cream
  Interventions: Dietary Supplement: Delivra TM Livsport preworkout cream; Dietary Supplement: Placebo
- LO Delivra TM Livsport preworkout cream (Experimental): 3.5 mL topical creatine + 3.5 mL placebo cream
  Interventions: Dietary Supplement: Delivra TM Livsport preworkout cream; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Delivra TM Livsport preworkout cream — High versus low dose topical creatine
Dietary Supplement: Placebo — Topical placebo

SUMMARY:
Creatine is a nutritional supplement that is often ingested to improve exercise performance. The advent of a new product that is applied to the skin overlying muscle offers potential benefit, if the creatine can be targeted to specific muscles. The investigators are testing a novel creatine cream to determine the effects on human muscular performance. The investigators are assessing the acute application of two different doses of the creatine cream on muscular power (determined by knee extension).

DETAILED DESCRIPTION:
Creatine monohydrate is a popular nutritional supplement with athletes involved in sports involving strength and power. When creatine is orally ingested it combines with inorganic phosphate to form phorylcreatine (PCr) in skeletal muscle . Adenosine Triphosphate (ATP) is the immediate source of energy in muscle - during exercise ATP is broken down to Adenosine Diphosphate (ADP) and inorganic phosphate. Duration of high-intensity exercise is limited to a few seconds based on limited ATP stores in muscle. PCr acts to re-phosphorylate ADP to form ATP so that muscle contraction can continue at high intensities. After creatine monohydrate is ingested, high-intensity exercise capacity is increased because of the increased PCr stores in muscle.

Delivra Inc. has developed a topical cream containing creatine that is designed to penetrate the skin. The study purpose is to determine whether the topical cream, at two different doses, is effective for improving muscular strength and power.

The hypotheses are that the experimental topical creatine cream will be more effective than a placebo cream for improving muscular performance and that two consecutive applications of creatine cream is more effective than a single application for improving muscular performance.

The study involves a involves a double-blind placebo-controlled parallel group design. Participants (n=132) will be randomized to receive either a low dose (3.5 mL) or high dose (7 mL) of topical creatine.

The baseline assessment involves measuring muscular power during 5 sets of 15 repetitions of knee extension on a dynamometer, with each set separated by 1 minute rest, with each leg tested separately. At least 72 hours after the baseline testing, participants will receive either a high or low dose of the topical creatine cream applied to the quadriceps of one leg. The high-dose group will receive 3.5 mL of creatine cream 30 minutes and 15 minutes to one leg (randomized) before exercise testing (i.e. the same testing as performed in visit 2). They will receive 3.5 mL of placebo cream 30 and 15 minutes to the opposite leg before testing. The low-dose group will receive placebo cream 30 minutes before testing and creatine cream 15 minutes before testing to one leg; they will receive placebo cream 30 and 15 minutes before testing on the opposite leg. Testing on each leg will involve measuring muscular power during 5 sets of 15 repetitions of knee extension on the dynamometer, with each set separated by 1 minute rest.

The primary outcomes are average and peak power output.

ELIGIBILITY:
Inclusion Criteria:

* Physically active and able to pass Physical Activity Readiness Questionnaire

Exclusion Criteria:

* Allergies to any ingredients in the cream
* Answering "yes" to Physical Activity Readiness Questionnaire
* Currently pregnant or breastfeeding,
* Presence of significant medical disorder that would compromise the participant's safety to take part in the trial (eg: cancer, immunosuppressed)
* History of alcohol or drug abuse within the past year
* Anyone using recreational drugs
* Use of performance enhancing drugs or supplements within 2 months including caffeine and creatine in supplement form
* Currently using other topical agents for treatment of pain or inflammation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2016-10; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in average power across 5 set of 15 repetitions separated by 60s rest on an isokinetic dynamometer | Change from baseline to one week (i.e. after application of creatine cream)

SECONDARY OUTCOMES:
Adverse events recorded on adverse event forms | Changes from baseline to one week (i.e. after application of creatine cream)
Change in peak power across 5 set of 15 repetitions separated by 60s rest on an isokinetic dynamometer | Change from baseline to one week (i.e. after application of creatine cream)

CONTACTS AND LOCATIONS:
Overall Officials: David Baranowski, Ph.D., Study Director — Delivra, Inc.; Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan; Jamie Burr, Ph.D., Principal Investigator — University of Guelph; Travis Saunders, Ph.D., Principal Investigator — UPEI
Locations (3):
- Canada (3):
  - University of Guelph, Guelph, Ontario
  - University of Prince Edward Island, Charlottetown, Prince Edward Island
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No